CLINICAL TRIAL: NCT05434676
Title: Clinical Trial of The ShOckwave Medical Peripheral Lithoplasty® System Used to Treat Moderate and Severely CalcIfied FemOropopliteal Arteries in ChiNese Patients (SOLUTION Trial)
Brief Title: SOLUTION Trial in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genesis Medtech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GM-PI-CIP002
Record Dates: First submitted 2022-06-15; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Peripheral Arterial Disease; Calcifications Vascular
MeSH Terms: conditions — Peripheral Arterial Disease; Vascular Calcification

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IVL group (Experimental): Shockwave Medical Peripheral Intravascular Lithotripsy (IVL) System M5 or S4
  Interventions: Device: Shockwave Medical Peripheral Intravascular Lithotripsy (IVL) System M5 & S4

INTERVENTIONS:
Device: Shockwave Medical Peripheral Intravascular Lithotripsy (IVL) System M5 & S4 — To assess the safety and effectiveness of IVL treatment used in combination with DCB to treat moderate and severely calcified femoropopliteal arteries

SUMMARY:
This is a prospective, multicenter, single arm study, to support the safety and effectiveness assessment of the Shockwave Medical Peripheral IVL System applied to Chinese patients

ELIGIBILITY:
Inclusion Criteria:

General

1. Subject or subject's legal representative have been informed of the nature of the study, agrees to participate and has signed the approved consent form.
2. Age of subject is > 18 and ≤80, male or female.
3. Rutherford Category 2 to 5 of the target limb (If both limbs are eligible for the study, one limb will be selected as the target limb at the discretion of the investigator)
4. Estimated life expectancy >1 year.
5. Subject is a suitable candidate for angiography and endovascular intervention in the opinion of the investigator or per hospital guideline.
6. Subject is intended to undergo treatment with IVL followed by DCB. Angiographic
7. Target lesion that is located in a native, de novo superficial femoral artery (SFA) or popliteal artery
8. Target lesion reference vessel diameter is between 4.0mm and 7.0mm by visual estimate.
9. Target lesion is ≥70% stenosis by investigator via visual estimate.
10. Target lesion length is ≤180mm for lesions 70-99% stenosed. Target lesion can be all or part of the 180mm treated zone.
11. Chronic total occlusion (CTO), lesion length is ≤100mm of the total ≤180mm target lesion.
12. Subject has at least one patent tibial vessel on the target leg with runoff to the foot, defined as no stenosis >50%.
13. Calcification is at least moderate defined as presence of fluoroscopic evidence of calcification: 1) on parallel sides of the vessel and 2) extending > 50% the length of the lesion if lesion is ≥50mm in length; or extending for minimum of 20mm if lesion is <50mm in length.

Exclusion Criteria:

General

1. Subject has active infection requiring antibiotic therapy.
2. Planned target limb major amputation (above the ankle).
3. History of prior endovascular or surgical procedure on the index limb within the past 30 days or planned within 30 days of the index procedure.
4. Subject has a known coagulopathy or has bleeding diatheses, thrombocytopenia with platelet count less than 100,000/microliter.
5. Subject in whom antiplatelet or anticoagulant therapy is contraindicated.
6. Subject has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
7. Subject has known allergy to urethane, nylon, or silicone.
8. Myocardial infarction within 60 days prior to enrollment.
9. History of stroke within 60 days prior to enrollment.
10. History of thrombolytic therapy within two weeks of enrollment.
11. Serum creatinine greater than 2 times the upper reference limit
12. Subject is pregnant or nursing.
13. Women of childbearing potential (18 years to less than 2 years post-menopausal and not surgically sterile) with positive blood or urine pregnancy test at screening
14. Subject is participating in another research study that has not reached the primary endpoint.
15. Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post- treatment.
16. The use of specialty balloons (Scoring or cutting balloon), re-entry or atherectomy devices.

    Angiographic
17. In-stent restenosis within 10mm of the target zone.
18. Lesions within 10mm of the ostium of the SFA or within 10mm of the ostium of the anterior tibial artery.
19. Evidence of aneurysm or thrombus in target vessel.
20. No calcium or mild calcium in the target lesion.
21. Target lesion within native or synthetic vessel grafts.
22. Subject has significant non-target lesion (>50% stenosis or occlusion) within target limb (e.g. iliac or common femoral) not successfully treated prior to treatment of the target lesion.
23. Subject requires treatment of a peripheral lesion on the ipsilateral limb distal to target site at the time of the index procedure.
24. Failure to successfully cross the guidewire across the target lesion; successful crossing defined as tip of the guidewire distal to the target lesion in the absence of flow limiting dissections or perforations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Procedural success | Immediately post index procedure
  defined as residual stenosis ≤30% without flow-limiting dissection (≥ grade D) post IVL treatment (prior to DCB)by angiographic core lab
Major Adverse Event (MAE) at 30 days | 30 days post index procedure
  defined as:
  * Need for emergency surgical revascularization of target limb
  * Unplanned target limb major amputation (above the ankle)
  * Symptomatic thrombus or distal emboli that require surgical, mechanical or pharmacologic means to improve flow and extend hospitalization
  * Perforations that require an intervention, including bail-out stenting

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Affilated Hanzhou First People's Hospital, Zhejiang University School of Medicine, Shanghai
  - Huashan Hospital, Shanghai
  - Shanghai Jiaotong university school of medicine，Renji Hospital, Shanghai
  - Shanghai Jiaotong University School of Medicine，The Ninth People's Hospital, Shanghai
  - Zhongshan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No